CLINICAL TRIAL: NCT03905408
Title: PLeurodesis Using Hypertonic Glucose Administration to Treat Post-operative Air Leaks Following Lung Resection Surgery (PLUG-I): Phase 1
Brief Title: Pleurodesis Using Hypertonic Glucose to Treat Post-operative Air Leaks
Acronym: PLUG-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard Malthaner, MD, Chair/Chief Thoracic Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLUG-I
Record Dates: First submitted 2019-03-26; First posted 2019-04-05 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Air Leak
Keywords: glucose; lung surgery; air leak; postoperative
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Escalating dose:
  Arm 1: 50 mL dextrose 50% Arm 2: 100 mL dextrose 50% Arm 3: 150 mL dextrose 50% Arm 4:, 200 mL dextrose 50%
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 50 mL Dextrose (Experimental): 50 mL of 50% dextrose
  Interventions: Drug: 50 mL of 50% Glucose
- 100 mL Dextrose (Experimental): 100 mL of 50% dextrose
  Interventions: Drug: 100 mL of 50% Glucose
- 150 mL Dextrose (Experimental): 150 mL of 50% dextrose
  Interventions: Drug: 150 mL of 50% Glucose
- 200 mL Dextrose (Experimental): 200 mL of 50% dextrose
  Interventions: Drug: 200 mL of 50% Glucose

INTERVENTIONS:
Drug: 50 mL of 50% Glucose — 1st dose
  Other Names: Dextrose
  Arms: 50 mL Dextrose
Drug: 100 mL of 50% Glucose — 2nd dose
  Other Names: Dextrose
  Arms: 100 mL Dextrose
Drug: 150 mL of 50% Glucose — 3rd dose
  Other Names: Dextrose
  Arms: 150 mL Dextrose
Drug: 200 mL of 50% Glucose — 4th dose
  Other Names: Dextrose
  Arms: 200 mL Dextrose

SUMMARY:
The investigators will define the most appropriate safe dose of D50 to heal air leaks in patients that have undergone lung resection surgery

DETAILED DESCRIPTION:
The investigators will define the most appropriate safe dose of D50 to heal air leaks in patients that have undergone lung resection surgery (Phase I study). Air leaks from unhealed lung tissue are one of the most common complications after lung surgery including wedge resection, segmentectomy and lobectomy. Air leaks can lead to a delay in chest tube removal, prolonged pain, increased infections, prolonged hospital stay, and increased costs to the health care system. Different agents have been used to heal air leaks by creating a pleurodesis (adhesions to obliterate the pleural space between the visceral and parietal pleura). The success with these agents has been variable and come with the cost of complications that have restricted their use the post-operative period. There has been recent interest in the use of 50% hypertonic glucose (D50) to create pleurodesis with encouraging reports coming mostly from Asia. The investigators have performed a pilot study using 180 mL of D50 instilled through the chest tube for the management of post lobectomy air leak with very encouraging results. This preliminary study used strict inclusion criteria of only lobectomy patients and excluded all patients with known diabetes or any postoperative hyperglycemia. It is unknown if these patients would have benefitted from D50. Also, the optimal dose of D50 was chosen empirically and never clearly defined by previous work. It has been reported that high doses of D50 have been associated with acute lung injury. It is therefore critical that the optimal safe dose is clarified.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Lung resection is a wedge, segmentectomy, lobectomy or bilobectomy
3. Procedure performed by video-assisted thoracic surgery (VATS) or by Thoracotomy
4. Presence of an air leak on the digital draining system on postoperative day 2

Exclusion Criteria:

1. Large air leak arbitrarily defined as more than 1000 mL/min
2. Allergy to local anesthetics
3. Hemodynamic instability
4. Untreated coronary artery disease
5. Need for respiratory support
6. Any other early post-operative complication
7. Immunity disorder
8. Large pleural fluid output empirically defined as more than 500 mL in the last 12 hours
9. Inability to give consent
10. Fasting glucose ≥ 14 mmol/L the morning of the intervention (arbitrarily chosen cut-off in which patients' diabetes is considered very poorly controlled)
11. Endocrinology service not available to co-manage patients with either diabetes, or a fasting blood glucose ≥ 7 mmol/L, or HbA1c > 6.5%
12. Postoperative evidence of an active thoracic (lung or pleura) infection with systemic inflammatory response syndrome (2 or more of temperature > 38, heart rate > 90, respiratory rate > 20, white blood cell count > 12)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events | 1 year
  occurrence of treatment related adverse events (Grade 3 and more as assessed to the CTCAE v4.0) at any given dose of D50

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No